CLINICAL TRIAL: NCT05081843
Title: Tobacco Initiation Prevention for Pittsburgh and Rural Area High School Students
Brief Title: Pittsburgh and Rural Area High School Tobacco Prevention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Jaime Sidani, Associate Professor, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY21030093; K12DA050607 (NIH)
Record Dates: First submitted 2021-10-04; First posted 2021-10-18 (Actual); Results first posted 2025-06-04 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Adolescent Behavior; Tobacco Use; E-Cig Use
MeSH Terms: conditions — Adolescent Behavior; Tobacco Use; Vaping

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Health Education Curriculum (Active Comparator): Students will receive the school's usual health education curriculum.
  Interventions: Behavioral: Usual health education curriculum
- Usual Health Education Curriculum plus Intervention (Experimental): Students will receive the school's usual health education curriculum. Students will also receive the intervention. Delivery of the intervention (i.e., timing, frequency) will be determined by discussing the results of the Aim 1 focus groups with teachers and administrators.
  Interventions: Behavioral: AD IT UP media literacy intervention; Behavioral: Usual health education curriculum

INTERVENTIONS:
Behavioral: AD IT UP media literacy intervention — AD IT UP was originally developed in 2006 as a classroom-based cigarette prevention program focused on traditional media influences, and was converted to a web-based program in 2011. In 2019, the AD IT UP program was updated substantially to include other forms of tobacco, such as e-cigarettes, and other forms of media, such as social media.
  Arms: Usual Health Education Curriculum plus Intervention
Behavioral: Usual health education curriculum — The schools' regular health education curriculum includes classroom lectures, hands on activities and group work.

SUMMARY:
This research project will explore the feasibility and acceptability of a web-based media literacy tobacco prevention program. The project will be conducted with 9th graders in two schools in the Pittsburgh area.

DETAILED DESCRIPTION:
Specific Aim 1: To assess 9th grade students' preferences for delivery of the web-based media literacy tobacco prevention program. Investigators will conduct focus groups with 9th grade students in each high school. Students will be shown clips from the program and asked to provide feedback about the preferred frequency and setting for the program.

Specific Aim 2: Investigators will conduct a pilot trial of the intervention via a cluster randomized controlled trial. The control group will receive their usual health education curriculum. The intervention group will receive their usual health education curriculum with the addition of the intervention. All students will be asked to complete a pre-test, a post-test, and two follow-up surveys (approximately 4 and 12 months post-intervention). Feasibility endpoints will include overall program completion, recruitment/attendance rates, and retention rates. Acceptability outcomes will assess student perceptions toward the intervention. A sub-aim will be to conduct focus groups and interviews with students, teachers, and administrators to assess implementation barriers and facilitators.

ELIGIBILITY:
Inclusion Criteria:

* 9th grade student
* enrolled at participating Pittsburgh-area school

Exclusion Criteria:

* Inability to read the surveys

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 318 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Sidani, PhD MPH, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Appropriate data from this project will be made available via the Open ScienceFramework, which is recommended by the University of Pittsburgh Library System.
  Shareable data generated during the project will include longitudinal survey results, which will contain both quantitative and qualitative information. Survey data will be sufficiently de-identified and formatted in a broadly accessible spreadsheet format. Generic participant ID numbers will be available to link data across survey timepoints. These data will be made available with accompanying metadata (i.e., file descriptors and codebook). For example, available codebooks will include labels and descriptors for each quantitative survey variable as well as definitions used for qualitative coding.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available approximately December 2023 and remain available for 3 years in accordance with the NIH Grants Policy Statement on Data Sharing.
Access Criteria: Interested researchers will contact the PI to request access.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Health Education Curriculum | Usual Health Education Curriculum Plus Intervention
Started | 158 | 160
Completed | 23 | 15
Not Completed | 135 | 145
Not completed — Lost to Follow-up | 135 | 145

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Health Education Curriculum | Usual Health Education Curriculum Plus Intervention | Total
Number analyzed (Participants) | 158 | 160 | 318
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 158 | 160 | 318
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: In one of our two schools, the administration did not want us to ask any questions about sex or gender. Therefore, this data reflects only the school that allowed this item.
  Participants
    number analyzed (Participants) | 26 | 21 | 47
    Female | 13 | 7 | 20
    Male | 13 | 14 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White, non-Hispanic | 97 | 109 | 206
  Black, non-Hispanic | 8 | 4 | 12
  Asian, non-Hispanic | 19 | 17 | 36
  Hispanic or Latino | 5 | 9 | 14
  American Indian/Alaskan Native, non-Hispanic | 6 | 3 | 9
  Multiracial, non-Hispanic | 4 | 3 | 7
  Other | 1 | 1 | 2
  Missing | 18 | 14 | 32
Region of Enrollment [Number; unit: participants]
  United States | 158 | 160 | 318
Susceptible to cigarette use [Count of Participants; unit: Participants] — Item asked: If one of your best friends offered you a cigarette, would you smoke it?
  Responses: Definitely Yes, Probably Yes, Probably No, Definitely No
  Susceptible if: answers anything other than Definitely No
  Participants
    Susceptible | 11 | 18 | 29
    Not Susceptible | 120 | 116 | 236
    Missing | 27 | 26 | 53
Susceptible to cigar smoking [Count of Participants; unit: Participants] — Item asked: If one of your best friends offered you a cigar, would you smoke it?
  Responses: Definitely Yes, Probably Yes, Probably No, Definitely No
  Susceptible if: answers anything other than Definitely No
  Participants
    Susceptible | 8 | 16 | 24
    Not Susceptible | 124 | 119 | 243
    Missing | 26 | 25 | 51
Susceptible to e-cigarette use [Count of Participants; unit: Participants] — Item asked: If one of your best friends offered you an e-cigarette, would you use it?
  Responses: Definitely Yes, Probably Yes, Probably No, Definitely No
  Susceptible if: answers anything other than Definitely No
  Participants
    Susceptible | 15 | 29 | 44
    Not Susceptible | 115 | 105 | 220
    Missing | 28 | 26 | 54
Susceptible to hookah use [Count of Participants; unit: Participants] — Item asked: If one of your best friends offered you a hookah, would you smoke it?
  Responses: Definitely Yes, Probably Yes, Probably No, Definitely No
  Susceptible if: answers anything other than Definitely No
  Participants
    Susceptible | 10 | 14 | 24
    Not Susceptible | 121 | 120 | 241
    Missing | 27 | 26 | 53
Attitudes toward tobacco products [Mean (Standard Deviation); unit: units on a scale] — Measure description: 9 items that assessed agreement with statements about nicotine and tobacco products (see Study Protocol and Statistical Analysis Plan for exact item wording).
  10-item response scale (Strongly Disagree -Strongly Agree) for each item; overall summary score calculated by averaging scores across all items. Higher score indicates worse outcome (i.e. more positive attitudes).
  units on a scale | 3.24 (1.53) | 3.32 (1.36) | 3.29 (1.45)
Normative Beliefs [Mean (Standard Deviation); unit: units on a scale] — Measure description: 6 items that assessed perceptions about friends' acceptance of NTPs (see Study Protocol and Statistical Analysis Plan for exact item wording).
  10-item response scale (Very Unacceptable -Very Acceptable) for each item; overall summary score calculated by averaging scores across all items. Higher score indicates worse outcome (i.e. more perception of friends' acceptance).
  units on a scale | 2.27 (1.63) | 2.14 (1.26) | 2.21 (1.46)
Tobacco media literacy [Mean (Standard Deviation); unit: units on a scale] — Measure description: 8 items adapted from the Smoking Media Literacy Scale (see Study Protocol and Statistical Analysis Plan for exact item wording).
  10-item response scale (Strongly Disagree -Strongly Agree) for each item; overall summary score calculated by averaging scores across all items. Higher score indicates worse outcome (i.e. less media literacy).
  units on a scale | 7.78 (1.69) | 7.79 (1.74) | 7.79 (1.71)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Eligible 9th Grade Students Recruited to Participate in the Study
Description: Parents will be asked to return an opt out form if they do not want their student to participate. Students will provide assent if they wish to participate. Recruitment will be determined by calculating the percentage of eligible 9th grade students not opted out by their parents that also provide assent.
Time Frame: 1 month
Population: These numbers are the number of students that were present in the classroom on the day of the initial data collection, and thus eligible to participate.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Health Education Curriculum | Usual Health Education Curriculum Plus Intervention
Number analyzed (Participants) | 218 | 194
Participants | 158 | 160

2. Primary Outcome: Percentage of Participants Retained Through the Final Data Collection
Description: Retention will be calculated as the percentage of 9th grade students who completed the baseline survey and also completed the 12 month follow-up survey.
Time Frame: 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Health Education Curriculum | Usual Health Education Curriculum Plus Intervention
Number analyzed (Participants) | 158 | 160
Participants | 23 | 15

3. Primary Outcome: Percentage of Participants Indicating Moderate to High Acceptability of the AD IT UP Program
Description: Acceptability of the intervention will be assessed with closed-ended and open-ended items on the post-test survey immediately following completion of the intervention.
  Students will be asked on a 5-point Likert scale with responses ranging from Strongly Agree to Strongly Disagree (with a neutral middle) their agreement about the following: "I enjoyed AD IT UP," "I understood AD IT UP," "AD IT UP was easy to use," "I tried my hardest when I was doing AD IT UP," "I think AD IT UP would be helpful to other kids my age," "I would recommend AD IT UP to a friend," and "I agree with AD IT UP's message." An answer of "Strongly Agree" or "Agree" on these items indicates high and moderate acceptability, respectively. Each of these items will be assessed individually, not as an overall scale.
  Open-ended items will ask: what the student would change about AD IT UP, what the student liked about AD IT UP, what made AD IT UP fun, and what made AD IT UP not fun.
Time Frame: post-test immediately following completion of the intervention
Population: This data is from the intervention students who completed the post-test only.
Measure: Count of Participants; unit: Participants
Arm/Group | Usual Health Education Curriculum Plus Intervention
Number analyzed (Participants) | 111
Participants
  Agreed with "I understood AD IT UP" | 81
  Agreed with "AD IT UP was easy to use" | 62
  Agreed with "I tried my hardest when using AD IT UP" | 66
  Agreed with "UP would be helpful to other kids my age" | 64
  Agreed with "I agree with AD IT UP's message" | 82

4. Secondary Outcome: Changes in Intention to Use Tobacco Products
Description: Items used in this analysis:
  If one of your best friends offered you a [NTP], would you smoke/use it?
  This item was repeated for cigarettes, hookah, e-cigarettes, and cigars/cigarillos.
  This item included the a 4-item response scale ranging from Definitely No to Definitely Yes for each of the 4 NTPs.
  Susceptibility was considered any response except "Definitely No" and totaled for a possible range of 0 to 4. Answering anything other than "Definitely No" on any item is considered susceptible to using tobacco products. These were totaled for a possible range of 0 to 4, with higher scores representing greater susceptibility.
Time Frame: baseline vs. 12 month follow-up
Population: NOTE: The original analysis was to be conducted for change between baseline and 12-month follow-up. Due to loss to follow-up over the 12-month tme period, the results presented here are for the immediate post-test, for which there was less loss to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Health Education Curriculum | Usual Health Education Curriculum Plus Intervention
Number analyzed (Participants) | 70 | 93
units on a scale | 0.386 (0.997) | 0.419 (1.116)
Statistical Analysis 1: Comparison: Usual Health Education Curriculum vs Usual Health Education Curriculum Plus Intervention; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.233, 95% CI 2-sided [-0.056 to 0.522]

5. Secondary Outcome: Changes in Attitudes Toward Tobacco Products
Description: Items to measure attitudes toward tobacco products will be included in all 4 surveys. These items include the following with a 10-item response scale ranging from Strongly Disagree to Strongly Agree.
  E-cigarettes are not as bad for your health as other products. Using tobacco products at parties is fun. (added: Using e-cigarettes at parties is fun) Tobacco products help you deal with problems or stress. Smoking helps people stay thin. People who use e-cigarettes are more fun to be around than people who don't use e-cigarettes.
  If someone starts using tobacco products every day, it is very hard for them to stop (reverse coded).
  Smoking makes a person look more attractive. It would be very easy for me to get e-cigarettes if I wanted them.
  Change in attitudes will be determined by the average increase or decrease in agreement with these items. These items will be assessed individually and as an overall scale (range 0-90, with higher scores indicating a worse outcome).
Time Frame: baseline vs. 12 month follow-up
Population: NOTE: The original analysis was to be conducted for change between baseline and 12- month follow-up. Due to loss to follow-up over the 12 month time period, the results presented here are for the immediate post-test, for which there was less loss to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Health Education Curriculum | Usual Health Education Curriculum Plus Intervention
Number analyzed (Participants) | 73 | 98
units on a scale | 3.09 (1.98) | 2.91 (1.25)
Statistical Analysis 1: Comparison: Usual Health Education Curriculum vs Usual Health Education Curriculum Plus Intervention; Test type: Superiority; p = 0.05, t-test, 2 sided; Median Difference (Final Values) = 0.534, 95% CI 2-sided [0.078 to 0.990]

6. Secondary Outcome: Changes in Normative Beliefs About Tobacco Products
Description: Items to measure normative beliefs about tobacco products will be included in all 4 surveys. These items ask participants their rate how acceptable the following statements are among their friends using a 10-item response scale ranging from Very Acceptable to Very Unacceptable:
  It is OK for people your age to smoke cigarettes. It is OK for people your age to use e-cigarettes. It is OK for people your age to use hookahs. It is OK for people your age to smoke cigars or cigarillos. A wealthy person is more likely to use tobacco products than a poor person. A successful person is more likely to use tobacco products than an unsuccessful person.
  Changes in normative beliefs will be determined by the average increase or decrease in perceived acceptability of these statements. These items will be assessed individually, as well as an overall scale (range 0-60 with higher scores indicating a worse outcome).
Time Frame: baseline vs. 12 month follow-up
Population: NOTE: The original analysis was to be conducted for change between baseline and 12-month follow-up. Due to loss to follow-up over the 12 month time period, the results presented here are for the immediate post-test, for which there was less loss to sollow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Health Education Curriculum | Usual Health Education Curriculum Plus Intervention
Number analyzed (Participants) | 73 | 94
units on a scale | 2.43 (2.07) | 2.25 (1.29)
Statistical Analysis 1: Comparison: Usual Health Education Curriculum vs Usual Health Education Curriculum Plus Intervention; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.326, 95% CI 2-sided [-0.177 to 0.829]

7. Secondary Outcome: Change in Tobacco-related Media Literacy
Description: Items to measure tobacco-related media literacy will be adapted from the Smoking Media Literacy Scale and included in all 4 surveys. The response scale for these 8 items is a 10-item scale from "Strongly Disagree" to "Strongly Agree."
  Changes in media literacy will be determined by the average increase or decrease in agreement with these items. These items will be assessed individually, as well as an overall scale (range 0-80, with higher scores indicating a worse outcome).
Time Frame: baseline vs. 12 month follow-up
Population: NOTE: The original analysis was to be conducted for change between baseline and 12-month followup. Due to loss to follow-up over the 12 month time period, the results presented here are for the immediate post-test, for which there was less loss to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Usual Health Education Curriculum | Usual Health Education Curriculum Plus Intervention
Number analyzed (Participants) | 74 | 100
units on a scale | 7.98 (1.68) | 8.89 (1.79)
Statistical Analysis 1: Comparison: Usual Health Education Curriculum vs Usual Health Education Curriculum Plus Intervention; Test type: Superiority; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 0.756, 95% CI 2-sided [0.208 to 1.31]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Usual Health Education Curriculum | Usual Health Education Curriculum Plus Intervention
All-Cause Mortality (participants affected / at risk) | 0/158 | 0/160
Serious Adverse Events (participants affected / at risk) | 0/158 | 0/160
Other Adverse Events (participants affected / at risk) | 0/158 | 0/160

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-16): https://cdn.clinicaltrials.gov/large-docs/43/NCT05081843/Prot_SAP_000.pdf